CLINICAL TRIAL: NCT01897103
Title: Platelet Activity in Vascular Surgery
Brief Title: Platelet Activity in Vascular Surgery for Thrombosis and Bleeding
Acronym: PIVOTAL
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Other Study IDs: 12-03123
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Peripheral Vascular Disease; Peripheral Artery Disease; Carotid Stenosis; Aortic Aneurysm, Abdominal; Aortic Aneurysm, Thoracic; Amputation, Wound; Embolism and Thrombosis; Aortic Aneurysm
Keywords: Peripheral Artery Disease; Endarterectomy (Carotid); Aortic Aneurysm, Abdominal; Aortic Aneurysm, Thoracic; Amputation; Platelet Activity; Thrombin; Transcriptomics
MeSH Terms: conditions — Peripheral Vascular Diseases; Peripheral Arterial Disease; Carotid Stenosis; Aortic Aneurysm, Abdominal; Aortic Aneurysm, Thoracic; Wounds and Injuries; Embolism and Thrombosis; Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, platelet RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The proposed PIVOTAL study will examine a panel of platelet/coagulation activity markers during the perioperative period. The goal is to develop a clinically useful assessment of platelet/coagulation activity for risk stratification that may ultimately serve as a target for therapeutic intervention. This study will enroll 200 patients with peripheral artery disease undergoing vascular surgery. PIVOTAL is funded by American Heart Association and is scheduled to begin enrollment in July 2013 for approximately two years.

DETAILED DESCRIPTION:
To describe platelet activity among PAD subjects undergoing vascular surgery.

To determine whether preoperative platelet activity measurements are independently associated with perioperative cardiovascular events.

To identify demographic, clinical, and surgical factors associated with postoperative platelet activity measurements in patients with established PAD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing non emergent vascular surgery
* Use of aspirin within 48 hours prior to surgery
* Age > 21 years of age
* Able and willing to provide written informed consent for the study

Exclusion Criteria:

* Use of any anticoagulant (Coumadin, heparin) within 24 hours to surgery
* Use of any Nonsteroidal Antiinflammatory Drug (NSAID) (such as ibuprofen, naproxen, etc.) within 72 hours
* Thrombocytopenia (platelet count<100) or Thrombocytosis (platelet count>500),
* Anemia (hemoglobin<9),
* Severe kidney disease (CrCl<30ml/min),
* Any known hemorrhagic diathesis.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population will be selected from the inpatient setting at NYU Medical Center and Bellevue Hospital as well as the outpatient setting in the Faculty Group Practice.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-06; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Platelet Activity | two years
  The main outcome measures are platelet activity, coagulation markers, platelet mapping and profiling.

SECONDARY OUTCOMES:
Perioperative Events | Two-years
  Thrombotic and Bleeding events

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Berger, MD, MS, FAHA, FACC, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - Bellevue Hospital Center, South Manhattan Healthcare Network, New York, New York
  - New York University School Of Medicine, New York, New York

REFERENCES:
- [Background] Berger JS, Hiatt WR. Medical therapy in peripheral artery disease. Circulation. 2012 Jul 24;126(4):491-500. doi: 10.1161/CIRCULATIONAHA.111.033886. No abstract available. PMID 22825411
- [Background] Berger JS, Becker RC, Kuhn C, Helms MJ, Ortel TL, Williams R. Hyperreactive platelet phenotypes: relationship to altered serotonin transporter number, transport kinetics and intrinsic response to adrenergic co-stimulation. Thromb Haemost. 2013 Jan;109(1):85-92. doi: 10.1160/TH12-03-0202. Epub 2012 Dec 6. PMID 23223800
- [Background] Chu SG, Becker RC, Berger PB, Bhatt DL, Eikelboom JW, Konkle B, Mohler ER, Reilly MP, Berger JS. Mean platelet volume as a predictor of cardiovascular risk: a systematic review and meta-analysis. J Thromb Haemost. 2010 Jan;8(1):148-56. doi: 10.1111/j.1538-7836.2009.03584.x. Epub 2009 Aug 19. PMID 19691485
- [Background] Eraso LH, Fukaya E, Mohler ER 3rd, Xie D, Sha D, Berger JS. Peripheral arterial disease, prevalence and cumulative risk factor profile analysis. Eur J Prev Cardiol. 2014 Jun;21(6):704-11. doi: 10.1177/2047487312452968. Epub 2012 Jun 27. PMID 22739687
- [Background] Sharma G, Berger JS. Platelet activity and cardiovascular risk in apparently healthy individuals: a review of the data. J Thromb Thrombolysis. 2011 Aug;32(2):201-8. doi: 10.1007/s11239-011-0590-9. PMID 21562837
- [Derived] Dann R, Hadi T, Montenont E, Boytard L, Alebrahim D, Feinstein J, Allen N, Simon R, Barone K, Uryu K, Guo Y, Rockman C, Ramkhelawon B, Berger JS. Platelet-Derived MRP-14 Induces Monocyte Activation in Patients With Symptomatic Peripheral Artery Disease. J Am Coll Cardiol. 2018 Jan 2;71(1):53-65. doi: 10.1016/j.jacc.2017.10.072. PMID 29301628